CLINICAL TRIAL: NCT04170608
Title: PEFCAT II: Expanded Safety and Feasibility Study of the FARAPULSE Endocardial Multi Ablation System to Treat Paroxysmal Atrial Fibrillation
Brief Title: PEFCATII Expanded Safety and Feasibility Study of the FARAPULSE Endocardial Multi Ablation System to Treat Paroxysmal Atrial Fibrillation
Acronym: PEFCATII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0571
Record Dates: First submitted 2019-10-17; First posted 2019-11-20 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- FARAPULSE Endocardial Ablation (Experimental): Ablation using the FARAPULSE Endocardial Multi Ablation System
  Interventions: Device: FARAPULSE Endocardial Multi Ablation System

INTERVENTIONS:
Device: FARAPULSE Endocardial Multi Ablation System — Ablation using the FARAPULSE Endocardial Multi Ablation System

SUMMARY:
PEFCAT II: Expanded Safety and Feasibility Study of the FARAPULSE Endocardial Multi Ablation System to Treat Paroxysmal Atrial Fibrillation

DETAILED DESCRIPTION:
This is a prospective, multi-center, safety and feasibility study. Subjects will undergo percutaneous PEF ablation for pulmonary vein isolation and at the clinical discretion of the investigator receive PEF ablation of additional arrhythmogenic locations. Subjects will be followed at 30 days, 75 days, 6 months and 12 months for adverse events, recurrence of arrhythmia after a 90-day Blanking Period and other relevant outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Study subjects are required to meet all the following inclusion criteria to participate in this study:

1. Patients with documented drug-resistant symptomatic PAF meeting all three of the following criteria:

   1. Confirmed AF: Documentation must include a recording such as ECG, transtelephonic monitor (TTM), Holter monitor, implanted devices, or telemetry strip, recorded within one year prior to enrollment and showing at least 30 seconds of AF.
   2. Frequent AF, defined as ≥ 2 episodes within 6 months of enrollment.
   3. Failed atrial fibrillation drug (AFD) treatment, meaning therapeutic failure of at least one AFD (class I - IV) for efficacy and / or intolerance.
2. Patients who are ≥ 18 and ≤ 75 years of age on the day of enrollment.
3. Patient participation requirements:

   1. Lives locally.
   2. Is willing and capable of providing Informed Consent to undergo study procedures.
   3. Is willing to participate in all examinations and follow-up visits and tests associated with this clinical study.

Exclusion Criteria:

EXCLUSION CRITERIA: Subjects will be excluded from participating in this study if they meet any one of the following exclusion criteria:

1. Atrial fibrillation that is any of the following:

   1. Persistent (by diagnosis or duration > 7 days)
   2. Secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible / non-cardiac causes
   3. Requires ≥ 4 cardioversions in the preceding 12 months
2. Left atrial anteroposterior diameter ≥ 5.0 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT)
3. Any of the following cardiac procedures, implants or conditions:

   1. Clinically significant arrhythmias other than AF, AFL or AT
   2. Hemodynamically significant valvular disease
   3. Prosthetic heart valve
   4. NYHA Class III or IV CHF
   5. Previous endocardial or epicardial ablation or surgery for AF
   6. Atrial or ventricular septal defect closure
   7. Atrial myxoma
   8. Left atrial appendage device or occlusion
   9. Pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices
   10. Significant or symptomatic hypotension
   11. Bradycardia or chronotropic incompetence
   12. History of pericarditis
   13. History of rheumatic fever
   14. History of congenital heart disease with any residual anatomic or conduction abnormality
4. Any of the following within 3 months of enrollment:

   1. Myocardial infarction
   2. Unstable angina
   3. Percutaneous coronary intervention
   4. Heart surgery (e.g. coronary artery bypass grafting, ventriculotomy, atriotomy)
   5. Heart failure hospitalization
   6. Stroke or TIA
   7. Clinically significant bleeding
   8. Pericarditis or pericardial effusion
   9. Left atrial thrombus
5. History of blood clotting or bleeding abnormalities
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Contraindications to CT or MRI
8. Sensitivity to contrast media not controlled by premedication
9. Women of childbearing potential who are pregnant, lactating or not using birth control
10. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to:

    1. Body mass index (BMI) > 40
    2. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
    3. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
    4. Renal insufficiency with an estimated creatinine clearance < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
    5. Active malignancy or history of treated cancer within 24 months of enrollment
    6. Clinically significant gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
    7. Clinically significant infection
    8. Predicted life expectancy less than one year
11. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the protocol requirements.
12. Current or anticipated enrollment in any other clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, Principal Investigator — Nemocnice Na Homolce
Locations (2):
- University Hospital of Split, Split, Croatia
- Nemocnice Na Homolce, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 subjects consented and were treated.
Pre-assignment Details: A total of 10 patients were enrolled (signed informed consent) and 10 subjects were treated at two (2) sites in Europe.
Period: Overall Study
Arm/Group | FARAPULSE Endocardial Ablation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 5
  Croatia | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.9 (3.3)
Left Atrial Diameter [Mean (Standard Deviation); unit: cm] | 3.9 (0.4)
AF History (number of months) [Mean (Standard Deviation); unit: Months] | 20.98 (0.1)
LVEF % [Mean (Standard Deviation); unit: Percentage of Left ventricular ejection] | 61.9 (5.0)
CHA2DS2VASC [Mean (Standard Deviation); unit: units on a scale] — Tool used to predict the risk of ischemic stroke in patients with AF, which can help guide the decision to treat those patients with anticoagulants. Calculated by adding the number of risk factors: CHF, hypertension, age ≥ 75,diabetes, stroke/TIA/TE, vascular disease, age 65-74 years, and sex. Each risk factor adds a point to the risk score, except for Age ≥ 75 years and Stroke/TIA/TE, which both add 2 points. A score of 0 represents no additional risk factors. ESC guidelines considers a score of 1 to be moderate risk and a score ≥ 2 to be high risk. Range: 0 (lower risk) - 9 (higher risk).
  units on a scale | 1.8 (1.7)
Patient that failed any AntiArrhythmic Drugs [Count of Participants; unit: Participants] | 10
Smoking [Count of Participants; unit: Participants] | 1
Dyslipidemia [Count of Participants; unit: Participants] | 3
COPD [Count of Participants; unit: Participants] | 0
Pace Maker/Implantable Cardioverter Defibrillator [Count of Participants; unit: Participants] | 0
Unstable angina [Count of Participants; unit: Participants] | 0
NYHA Heart Failure Class I [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 0
NYHA Heart Failure Class II [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 3
NYHA Heart Failure Class III [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 0
NYHA Heart Failure Class IV [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 0
Any History of Structural heart disease [Count of Participants; unit: Participants] | 0
Cerebrovascular disease [Count of Participants; unit: Participants] | 1
Cardiac Surgery [Count of Participants; unit: Participants] | 0
Diabetes [Count of Participants; unit: Participants] | 1
Hypertension [Count of Participants; unit: Participants] | 6
Hyperthyroidism [Count of Participants; unit: Participants] | 0
Hypothyroidism [Count of Participants; unit: Participants] | 3
Myocardial infarction [Count of Participants; unit: Participants] | 0
Peripheral vascular disease [Count of Participants; unit: Participants] | 0
Pulmonary hypertension [Count of Participants; unit: Participants] | 0
Renal dysfunction/failure [Count of Participants; unit: Participants] | 1
Sleep apnea [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Prespecified Primary Safety Events Within 30 Days of Index Procedure.
Description: Number of patients with death, MI, diaphragmatic paralysis, stroke/TIA, thromboemolism, pericarditis, tamponade/perforation, vascular access complications, hospitalization, heart block, PV stenosis, atrioesophageal fistula.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 10
Participants | 0

2. Primary Outcome: Feasibility: Acute Key Procedural Success
Description: The primary feasibility endpoint for this study is the proportion of subjects that achieve Acute Procedural Success (APS) defined as the percutaneous endocardial creation of a complete, electrically isolating set of lesions around the ostia of the pulmonary veins (PVI) using the FARAPULSE Endocardial Multi Ablation System during the first Procedure, as clinically assessed by entrance and/or exit block performed ≥ 20 minutes after the last PVI lesion is made.
Time Frame: Index Procedure
Measure: Number; unit: Proportion of subjects
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 10
Proportion of subjects | 1.0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | FARAPULSE Endocardial Ablation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Endocardial Ablation (N=10)
Headache (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Injection site inflammation (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Disorders (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Blood and lymphatic system disorders) | 1 (1)
Sinus Arrest (Cardiac disorders) | 1 (1)
Gastrointestinal Tract Irritation (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04170608/Prot_SAP_000.pdf